CLINICAL TRIAL: NCT04890288
Title: aPneic oxygEnation duriNg emerGent intUbation of crItically Ill childreN: a Multi-center Randomized Controlled Trial
Brief Title: Apneic Intubation Critically Ill Children
Acronym: Penguin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Geneva (Other); State Hospital, St. Gallen (Other Government); University of Zurich (Other); Luzerner Kantonsspital (Other); Kantonsspital Graubuenden (Other); Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-02609
Record Dates: First submitted 2020-12-03; First posted 2021-05-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Airway Management
Keywords: Pediatric; Intubation; Apnea; Desaturation; High flow
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group - High flow (Experimental): High-flow nasal cannula oxygen 2L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0; enabling apneic oxygenation during laryngoscopy.
  Interventions: Procedure: Interventional randomized controled trial (RCT) comparing two oxygenation methods to reduce desaturation during intubation vs standard of care.
- Intervention group - Low flow: (Experimental): Low-flow oxygen (100%, 0.2 l/kg/min) via conventional neonatal nasal cannula (Intersurgical, Wokingham, Berkshire, United Kingdom) enabling apneic oxygenation during laryngoscopy.
  Interventions: Procedure: Interventional randomized controled trial (RCT) comparing two oxygenation methods to reduce desaturation during intubation vs standard of care.
- Conventional (No Intervention): Conventionally practiced standard of care with preoxygenation with facemask with an FiO2 of 1.0, followed by bag mask ventilation after induction before oral intubation without apneic oxygenation.

INTERVENTIONS:
Procedure: Interventional randomized controled trial (RCT) comparing two oxygenation methods to reduce desaturation during intubation vs standard of care. — Demonstrate that airway management supported by oxygen supplementation (either HFNC or low flow oxygen) can prevent significant desaturation (SpO2 > 85%) among patients in pediatric intensive care units (PICU) and neonatal intensive care units (NICU).
  Arms: Intervention group - High flow; Intervention group - Low flow:

SUMMARY:
This study compares the actual standard of care of intubation in Swiss pediatric intensive care units vs the use of apneic oxygenation using either high flow or low flow oxygen to prevent hypoxemia and to prolong apnea time during intubation of critically ill children, with the final aim to improve airway management safety at PICUs. Primary study objective: To demonstrate that airway management supported by oxygen supplementation (either HFNC or low flow oxygen) can prevent significant desaturation (SpO2 > 85%) among patients in pediatric intensive care units (PICU) and neonatal intensive care units (NICU).

DETAILED DESCRIPTION:
Randomized controlled multicenter trial in Swiss pediatric ICUs with randomization to 3 groups: 1) standard of care with conventional preoxygenation with bag-mask ventilation vs 2) conventional preoxygenation with bag-mask ventilation and apneic oxygenation with low-flow Oxygen fraction of inspired oxygen (FiO2) 100% 0.2 L/kg/min vs 3) conventional preoxygenation with bag-mask ventilation and apneic oxygenation with THRIVE FiO2 100% 2L/kg/min.

Eligible children meeting the inclusions criteria will be prepared for oral intubation according to the standard operating procedure (SOP) of the respective NICU/PICU. SpO2, heart rate, invasive or non-invasive blood pressure values shall be recorded continuously (for invasive continuously and for non-invasive intermittently every 2 minutes and 30 seconds), once the decision to intubate has been made. The sealed envelope for randomization will then be opened. All patients must be intubated orally. The induction will be performed according to the clinical needs of the child. All children will be intubated using the C-MAC videolaryngoscope with a Miller or Macintosh-blades (Karl Storz, Tuttlingen, Germany) age adopted.

Before oral intubation preoxygenation is performed for 2 minutes with a facemask usually used at the study site with an FiO2 of 1.0 and flow rates of 6-10L/min in all groups. After induction, all patients will be paralyzed with an age appropriate dose of muscle relaxant to ensure apnoea. The dose of the neuromuscular blocking agent and the depth of the anesthesia shall be adjusted according to clinical parameters such as absent reactions to jaw thrust and normocardia. In all groups, after induction, bag-mask ventilation with 100% oxygen and flow rates of 6-10 Lmin-1 will be continued for about 45-60 seconds until apnea sets in. Thereafter bag-mask ventilation will be stopped and one of the three study interventions will be applied according to randomization:

Control group: When apnea sets in, deep laryngoscopy and endotracheal oral intubation are performed without apneic oxygenation.

Intervention group - high flow: Prior to the introduction of the laryngoscope, apneic oxygenation is commenced with a high-flow nasal cannula flow rate of 2L/kg/min using OptiFlow system at an FiO2 of 1.0. After starting THRIVE laryngoscopy and tracheal oral intubation is performed.

Intervention group - low flow: Prior to the introduction of the laryngoscope, the administration of low-flow oxygen (0.2 l/kg/min) will take place via conventional neonatal nasal cannula (Intersurgical, Wokingham, Berkshire, United Kingdom). After starting low-flow oxygen laryngoscopy and tracheal oral intubation is performed.

A chest x-ray, which is a routine procedure, shall be performed at the conclusion of the procedure to verify the endotracheal tube (ETT) position and rule out a pneumothorax.

Study termination criteria constitute successful intubation or the occurrence of a "Can't Intubate, Can't Oxygenate" emergency. A maximum of 4 intubation attempts in total may be performed. The last intubation attempt must be performed by the most experienced physician in the room. Additional devices like stylet, bougie, etc, can be used at any stage of the intubation process. If the intubation remains unsuccessful the difficult airway algorithm will be followed and a supraglottic airway device (SAD) device will be inserted. Unsuccessful intubation requiring a SAD will lead to immediate study termination. Equipment malfunction (e.g. HFNC, C-MAC VL) will lead to study cessation. In the event of an unexpected difficult intubation, the difficult airway algorithm will be followed.

Intervention group - High flow: High-flow nasal cannula oxygen 2L/kg/min using OptiFlow system by Fisher&Paykel and an oxygen inspiration concentration FiO2 of 1.0; enabling apneic oxygenation during laryngoscopy.

Picture showing nasal prongs for high-flow oxygen. Intervention group - Low flow: Low-flow oxygen (100%, 0.2 l/kg/min) via conventional neonatal nasal cannula (Intersurgical, Wokingham, Berkshire, United Kingdom) enabling apneic oxygenation during laryngoscopy.

Conventionally practiced standard of care with preoxygenation with facemask with an FiO2 of 1.0, followed by bag mask ventilation after induction before oral intubation without apneic oxygenation.

The investigators will include 210 patients, 70 per group. Assuming a desaturation rate of 40% in the control group and a desaturation rate of max 15% with low-flow oxygen and HFNC, aiming at a power of 80% and setting an alpha-level at 0.025 the investigators would need n=56 patients per group. Accounting for some drop-outs, they seek to enroll n=70 patients per group, i.e. a total of n=210 patients.

In pilot studies to this protocol and in recent published data a maximum desaturation of 10% was observed during intubation for both therapies.

The difference in desaturation rate between the 2 intervention groups will be analyzed for non-inferiority.

Assuming a desaturation rate of 85% with HFNC and desaturation rate of 85 % with low-flow oxygen, aiming at a power of 80% and setting an alpha-level at 0.025 (one-sided non-inferiority trial), with a non-inferiority limit of 17% the investigators would need n=70 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring intubation in the pediatric intensive care unit
* Aged from 37 weeks corrected gestational age to 6 years
* Legal guardians providing written informed consent before the intervention or delayed consent in the event that emergency intubation is required

Exclusion Criteria:

* Patients with known or suspected difficult/airways
* Congenital heart disease mandating FiO2 < 1.0, warranting inhalational induction, requiring ongoing CPR or advanced life support due to respiratory arrest
* Preterm age < 37 0/7 weeks
* Patients who cannot be intubated orally
* Respiratory insufficiency with an SpO2 saturation < 90 % after 2 min of preoxygenation with FiO2 = 1.0
* Newborns requiring surfactant within the first 3 days of life
* Document stating intent to reject participation in research projects or refusal of intubation or refusal of resuscitation measures

Ages: 37 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with desaturation < 85 percent during intubation | 15 minutes
  To demonstrate that airway management supported by oxygen supplementation (either HFNC or low flow oxygen) can prevent significant desaturation (SpO2 > 85%) among patients in pediatric intensive care units (PICU) and neonatal intensive care units (NICU).

SECONDARY OUTCOMES:
Number of patients with desaturation low-flow oxygen vs. HFNC | 15 minutes
  Difference in desaturation between low-flow oxygen and HFNC
First attempt success rate | 15 minutes
  Rate of successful tube placement upon first attempt
Number of attempts | 15 minutes
  overall number of intubation attempts
Time required for intubation | 5 minutes
  Time required for intubation (in seconds), defined by the moment the laryngoscope passes the lips until successful lung ventilation is confirmed (defined as positive capnography)
Duration of desaturation < 85 percent | 15 minutes
  Duration of desaturation below 85%
Level of desaturation < 85 percent | 15 minutes
  Degree of desaturation below 85%

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Study Chair — University of Berne
Locations (7):
- Switzerland (7):
  - EOC, Bellinzona
  - Inselspital, Bern
  - Kantonsspital, Chur
  - HUG, Geneva
  - Kantonsspital Luzern, Lucerne
  - Kinderspital, Sankt Gallen
  - Kinderspital, Zurich

IPD SHARING:
Plan to Share IPD: No